CLINICAL TRIAL: NCT02891538
Title: A Pilot Study to Evaluate the Chemopreventive Effects of Epigallocatechin Gallate (EGCG) in Colorectal Cancer (CRC) Patients With Curative Resections.
Brief Title: Chemopreventive Effects of Epigallocatechin Gallate (EGCG) in Colorectal Cancer (CRC) Patients
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Sukeshi Patel, Principal Investigator, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CTMS 16-0085; 16-446H (Other: UT Health San Antonio)
Record Dates: First submitted 2016-08-31; First posted 2016-09-07 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-03

CONDITIONS: Colon Cancer
Keywords: EGCG; Green Tea; Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — epigallocatechin gallate; Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- epigallocatechin gallate (EGCG) (Experimental): Patients randomized to the EGCG arm, will start EGCG within 4-12 weeks of surgery and take EGCG 450 mg PO twice a day.
  Interventions: Drug: Epigallocatechin gallate (EGCG)
- Observation Only (No Intervention): Standard of care surgical resection followed by standard of care colonoscopy at year.

INTERVENTIONS:
Drug: Epigallocatechin gallate (EGCG) — Teavigo™ is a natural, caffeine-free, highly purified and refined green tea extract providing 94% epigallocatechin gallate (EGCG).*
  Other Names: Green Tea Extract
  Arms: epigallocatechin gallate (EGCG)

SUMMARY:
This will be a randomized, controlled pilot trial of patients with histological documentation of primary colon or rectal adenocarcinoma with resectable cancer, who have not received any treatments for cancer. If patient is a candidate for surgical resection, with no planned neoadjuvant chemotherapy, then the patient is eligible. All eligible subjects will be consented prior to surgery.

DETAILED DESCRIPTION:
Part 1: Blood draw prior to surgery, followed by surgical resection, and surgical pathologic specimen will be archived. After surgery, patient will be seen in 4-12 weeks to determine if adjuvant chemotherapy is indicated, in which case patient will receive adjuvant therapy. At this visit a blood draw will be done.

Part 2: If the patient is stage 0/1/2 and no plan for adjuvant treatments, then the patient will be randomized in a 2:1 manner to EGCG 900 mg daily vs observation (standard of care) for 1 year. Patients randomized to the EGCG arm, will start EGCG within 4-12 weeks of surgery and take EGCG 450 mg PO twice a day. Blood draw will be done at 0, 3, 6, 9, 12, 15, 18 months. Colonoscopy will be done at 1 year from diagnosis, at which time normal colonic tissue biopsies as well as any resected polyps will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically or histologically confirmed of primary colon or rectal adenocarcinoma with resectable cancer, who have not received any treatments for cancer.
* Age 18 years and above
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* The patient is a candidate for surgical resection, with no planned neoadjuvant chemotherapy, and there is a planned surgery for the primary colorectal cancer cancer or the patient had recent resection of the primary colorectal cancer. .
* For women who are not postmenopausal (12 months of amenorrhea) or surgically sterile (absence of ovaries and/or uterus): agreement to use two adequate methods of contraception. For men: agreement to use a barrier method of contraception during the treatment period
* Hematologic, Biochemical, and Organ Function within 7 days prior to Cycle 1 Day 1: Granulocyte count > 1000/mm3, Platelet count > 50,000/ mm3, Hemoglobin > 7 g/dL; Total bilirubin < 1.5xULN; Albumin > 2.8g/dl; aspartate aminotransferase (AST) (SGOT) and alanine aminotransferase (ALT) (SGPT) </=2.5 x upper limit of normal (ULN); Serum creatinine< 2 x ULN

Exclusion Criteria:

* Patients receiving prior chemotherapy or chemoradiation for colorectal cancer (ie, neoadjuvant chemoradiation for stage II or III rectal cancer).
* Known diagnosis of stage III colon or rectal cancer will be excluded from the study.
* Patients with metastatic disease.
* Patients may not be receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to green tea or EGCG.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease. Patients with nasogastric tube (NG-tube), J-tube, or G-tube will not be allowed to participate.
* Pregnant women are excluded from this study because of unknown effects of EGCG on teratogenic or abortifacient effects. For this reason, women of childbearing potential and men must also agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation.
* Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with EGCG, breastfeeding should be discontinued.
* Informed Consent - No study specific procedures will be performed without a written and signed informed consent document. Patients who do not demonstrate the ability to understand or the willingness to sign the written informed consent document will be excluded from study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2025-12-02 (Estimated)

PRIMARY OUTCOMES:
Change in methylation from baseline when compared to the control arm | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sukeshi Patel, MD, Principal Investigator — CTRC (Cancer Therapy and Research Center) at UTHSCSA
Locations (1):
- UT Health San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No